CLINICAL TRIAL: NCT06757842
Title: Acceptability and Feasibility of an 8-week In-person Mindfulness-Based Cognitive Therapy Program in a University Population: a Quasi-experimental Pilot Study
Brief Title: Acceptability and Feasibility of an In-person 8-week Mindfulness-Based Cognitive Therapy Program Among Undergraduates
Acronym: MFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Jorge Gaete, Full Professor, Universidad de los Andes, Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FDI UAN23102 - Mindfulness; FDI UAN23102 (Other Grant/Funding Number: Agencia Nacional de Investigacion y Desarrollo)
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Depression/Anxiety
Keywords: Depression; Anxiety; Undergraduates; Mindfulness
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental study without a control group, with pre- and post-intervention assessments. The intervention consists of an eight-week, in-person mindfulness training aimed at the university population
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The mindfulness intervention consists of eight group mindfulness skills sessions, held weekly in person at Universidad de los Andes, each lasting 90 minutes. The sessions will be co-facilitated by 2 instructors. One will lead the session activities, and the second facilitator will provide technical assistance for the session, monitor adverse events, and offer support to participants who may need it.
  Interventions: Behavioral: Mindfulness in Students

INTERVENTIONS:
Behavioral: Mindfulness in Students — The mindfulness intervention includes eight 90-minute group sessions held weekly at Universidad de los Andes, co-facilitated by two instructors. One leads the activities, while the other assists with technical aspects, monitors adverse events, and provides participant support. Participants will receive mindfulness worksheets and are required to practice at home for 15 minutes daily. They will have access to an online platform with audiovisual materials to guide their practice and will complete home practice logs online. Skills taught include sitting meditation (focused on breathing, thoughts, emotions, or sensations), body scan meditation, standing meditation, and mindfulness of daily activities. Group discussions will cover topics such as defining mindfulness, managing stress and pain, the difference between mindfulness and being on 'autopilot,' and how perceptions affect stress, as well as the relationship between pain and suffering, and the acceptance of unwanted experiences.

SUMMARY:
Mental health among university students has emerged as a significant global issue. Recent meta-analyses reveal that 25% of students experience depressive symptoms and 14% exhibit suicidal behaviors. A study involving 19 universities across 8 countries found that 31.4% reported psychiatric disorders in the past year, particularly major depressive episodes and anxiety disorders.

In Chile, research on university mental health is limited. A 2014 study at Universidad Austral reported a 27% prevalence of depression and a 5.3% risk of moderate to severe suicide risk. The "First National Survey of University Mental Health" in 2019 revealed that 46% of students had depressive symptoms, while health surveys from Universidad de los Andes in 2020 and 2022 showed a decrease in these symptoms, although suicide risk remained high.

Given this situation, preventive interventions are urgently needed. "Mindfulness-Based Interventions" (MBIs) have shown effectiveness in university settings. Mindfulness, defined by Jon Kabat-Zinn, involves deliberate, non-judgmental attention to the present moment. Programs like "Mindfulness-Based Stress Reduction" (MBSR) have proven effective in reducing symptoms of depression, anxiety, and stress. Studies indicate that MBIs can effectively alleviate mental health symptoms in university populations.

Some of the MBIs include "Mindful Mood Balance" (MMB) and "Mindfulness Skills for Students". The latter has shown effectiveness in reducing depressive and anxious symptoms among university students.

A 2021 pilot study at Universidad de los Andes on an online 8-session intervention combining mindfulness with cognitive-behavioral techniques yielded positive results in reducing symptoms and enhancing students' quality of life.

In the current proposal we want to evaluate the feasibility and acceptability of the "Mindfulness Skills for Students" program delivered in-person by two trained facilitators. Additionally, we want to explore the efficacy of this intervention in reducing depressive, anxious, and stress symptoms among undergraduate students at Universidad de los Andes, using a quasi-experimental study design.

DETAILED DESCRIPTION:
Mental health among university students has become a common and serious problem in higher education institutions worldwide in recent years. Over the past five years, various meta-analyses and systematic reviews have revealed concerning figures across the board. A recent meta-analysis found that the average prevalence of depression (from eight studies with 13,790 participants) was 25% (95% CI: 17%, 35%), and the combined prevalence of suicidal behaviors (from four studies with 2,586 participants) was 14% (95% CI: 0%, 44%). In another study that included 19 universities across eight countries (Australia, Belgium, Germany, Mexico, Northern Ireland, South Africa, Spain, and the U.S.) with responses from 13,984 students, it was found that the prevalence of any psychiatric disorder in the past 12 months was 31.4%. Among these disorders, the presence of a major depressive episode (18.5%), generalized anxiety disorder (16.7%), substance use disorder (3%), and alcohol use disorder (6.3%) were highlighted.

In Chile, there are very few studies addressing the prevalence of mental health disorders and associated risk factors in the university population. The article published in 2014 by Baader et al. is one of the first records we have in our country, conducted with a population of 800 students during 2008 at the Universidad Austral, reporting a prevalence of 27% for depression and 5.3% of students at moderate to severe risk of suicide. In April and May 2019, the results of the "First National Survey of University Mental Health" were presented, a project led by the Universidad Católica de Temuco and sponsored by the National Agency for Research and Development (ANID), conducted with 600 students from the Universidad Católica de Temuco, the Universidad de Concepción, and the Universidad de Tarapacá. This project showed that 46% of students exhibited depressive symptoms, 46% exhibited anxiety symptoms, and 53.5% exhibited stress symptoms. Furthermore, 29.7% presented all three symptoms simultaneously, and 5.1% of students had suicidal thoughts at the time of the study.

The data obtained from the Mental Health Surveys at the Universidad de los Andes, conducted in 2020 and 2022 among undergraduate students, indicate variations in the prevalence of different psychological symptoms and risks. Specifically, the prevalence of depressive symptoms decreased from 37.1% to 27.84%, while anxiety symptoms slightly reduced from 37.9% to 36.13%. Regarding stress, a notable decrease was observed, dropping from 54.6% to 12.9%. On the other hand, the prevalence of suicidal risk experienced a less pronounced decrease, from 20% to 18.4%, remaining at a considerably high index.

Given this situation, it is urgent to find preventive alternatives to address these issues. Among the interventions that have shown the most evidence in the last decade are "Mindfulness-Based Interventions" (MBI). This has prompted the incorporation of these interventions into the university setting. For example, by 2015, nearly 80% of the 140 accredited medical schools in the United States had incorporated some type of MBI into their curricula. Mindfulness refers to an intrinsic and modifiable capacity of the human mind, defined by Jon Kabat-Zinn as "the awareness (qualitative) that emerges when paying attention deliberately, in the present moment, and without judgment to experience moment to moment." Currently, there are various standardized therapeutic programs that teach skills based on mindfulness. The first one developed was the "Mindfulness-Based Stress Reduction" (MBSR), created by Jon Kabat-Zinn in the 1970s, who combined Buddhist meditation Dharma, psychological therapies, and advances in neuroscience, establishing the first milestone in the development of mindfulness as a health intervention, originally focused on alleviating symptoms in patients with chronic pain associated with systemic pathologies.

Subsequently, a group of behavioral therapists trained by Mark Williams, Zindel Segal, and John Teasdale created a program based on Jon Kabat-Zinn's model combined with cognitive-behavioral therapy, focused on preventing relapse in patients with major depressive disorder, called "Mindfulness-Based Cognitive Therapy (MBCT)." Both programs have a series of similarities and differences in their methodology. They are both based on mindfulness, but the fundamental difference is that MBCT focuses on identifying symptoms related to depression and anxiety, while MBSR focuses on identifying the effects of stress on the patient's life.

MBIs have been applied to various groups of patients with different health conditions and to healthy individuals, where studies have shown positive results in reducing depressive, stress, and anxiety symptoms, achieving mild to moderate benefits, both as monotherapy and as a complement to drug therapy. Within the university population, there are systematic reviews, meta-analyses, and clinical trials that show a correlation in the reduction of these symptoms. There have also been shortened interventions that have shown statistically significant benefits in students' symptoms.

Regarding the potential risks of MBIs, there is no high-quality evidence that definitively establishes the negative effects that mindfulness practice may entail for individuals. The most comprehensive study on this topic is a multicenter survey on the unexpected effects of meditation, conducted at various institutions between Spain and Brazil. Its results reflect that nearly 25% of participants reported experiencing some type of unexpected effect to varying degrees due to meditation practice, with between 1-4% reporting more severe effects. Among the most common complaints were the emergence or increased intensity of anxiety, pain, depression, and, to a much lesser extent, dissociative symptoms. However, none of these discomforts led practitioners to discontinue their meditation practice. Concerning expert opinions or case reports, it is relevant to highlight the precautions suggested by Zindel Segal, one of the creators of the MBCT program, which contraindicates the intervention in patients with acute psychiatric comorbidities, individuals with active suicidal ideation without treatment, and patients with untreated trauma.

Various adaptation protocols have been proposed, and one of the most notable is the one designed by Zindel Segal's group, one of the original authors of the MBCT program, called Mindful Mood Balance (MMB), which consists of a platform with audiovisual material (videos, audios, images, etc.) aimed at the self-application of the MBCT program. The effectiveness of this intervention has been studied in adult populations with anxious and depressive symptoms, demonstrating a significant decrease in PHQ-9 and General Anxiety Disorder-7 scores.

There is also a program crreated by Dr Elizabeth English and evaluated by Dr. Julieta Galante et al. in 2018, called "Mindfulness Skills for Students," applied in Cambridge, consisting of an abbreviated 8-week MBCT program. Unlike MMB, it includes guidance from mindfulness specialists to direct the practice and has the advantage of demonstrating positive results related to depressive and anxious symptoms in the university population. Thanks to a collaboration with Dr. Galante, we have been able to translate and adapt the "Mindfulness Skills for Students" program, which will be the basis for the intervention to be evaluated in this research project. In this regard, in 2021, a pilot study with a control group was conducted at the Universidad de los Andes (ClinicalTrials.gov Identifier: NCT05114824) that evaluated an online mindfulness-based intervention with cognitive-behavioral elements over 8 sessions among undergraduate students, showing a significant reduction in depressive and anxiety symptoms and an increase in quality of life among those who participated in the intervention compared to the control group. Another study in England evaluated a mindfulness intervention, which achieved notable reductions in perceived stress, anxiety, and depression compared to a control group, with sustained benefits during follow-ups at 3 and 6 months.

n the current proposal we want to evaluate the feasibility and acceptability of the "Mindfulness Skills for Students" program delivered in-person by two trained facilitators. Additionally, we want to explore the efficacy of this intervention in reducing depressive, anxious, and stress symptoms among undergraduate students at Universidad de los Andes, using a quasi-experimental study design.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students at the Universidad de los Andes.
* Aged 18 or older.
* Capable of reading and speaking Spanish.
* With a score on the PHQ-9 depression scale between 0 and 14.
* Have participated in an informational meeting about the study and the implications of the intervention.
* Availability to attend 1 weekly session of 90 minutes for 8 consecutive weeks, and time to practice mindfulness exercises at home for at least 15 minutes daily during the intervention period.

Exclusion Criteria:

* With a PHQ-9 score greater than or equal to 15.
* With active suicidality, defined as score ≥ 3 in Columbia suicide severity scale.
* Currently undergoing psychiatric treatment for a severe condition, understood as: psychotic disorders and/or substance abuse.
* History of hospitalization for psychiatric conditions in the last 2 years.
* History of having participated in a previous MBI course, such as: MBCT, MBSR, MMB, among others.
* History of sexual abuse in their lifetime.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability Assessment | through study completion, an average of 2 year
  Acceptability will be evaluated by determining how this intervention program is received by students and the extent to which this intervention relates to the needs of this target population. The research team will develop an acceptability and satisfaction questionnaire and apply it to the intervention students
Feasibility Assessment: Number of participants recruited | through study completion, an average of 2 year
  Initially, inclusion and exclusion criteria will be defined to ensure that participants are representatives of the target group. A tracking system will be implemented to monitor the number of people recruited.
Feasibility Assessment: Recruitment time for completion | through study completion, an average of 2 year
  A tracking system will be implemented to monitor the time needed to complete the recruitment process.
Feasibility Assessment: Evaluation of data collection and results. | through study completion, an average of 2 year
  Clear protocols will be established for data collection and analysis, ensuring accuracy and consistency. Statistical analyzes will be used to check the validity and reliability of the results.
Feasibility Assessment: Evaluation of the acceptability of the intervention | through study completion, an average of 2 year
  Surveys will be used to collect opinions and perceptions of participants about the intervention and the methods used.
Client Satisfaction Questionnaire (CSQ-8) | through study completion, an average of 2 year
  It is an 8-item instrument validated in English and translated and validated into Spanish that measures general satisfaction with health services received in various populations. The answers are Likert-type with four options each. In addition, there is space to write down comments and suggestions. This instrument will be slightly adapted to questions oriented to the study context. The Customer Satisfaction Questionnaire has an internal consistency ranging between α=0.83 and α=0.93.
  Each item on the CSQ-8 is rated on a 4-point scale, generally ranging from 1 (low satisfaction) to 4 (high satisfaction). Therefore, the minimum possible score on the CSQ-8 is 8 (1 point on each of the 8 items), and the maximum score is 32 (4 points on each item).
  A higher score on the CSQ-8 indicates greater client satisfaction with the services received, which is considered a better outcome. In this context, a higher score is better, as it reflects a better customer perception of the service.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | through study completion, an average of 2 year
  It is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which rates each of the 9 Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria from "0" (Never) to "3" (Almost Every Day). In Chile, it has been validated among people aged 20 years and over, with a sensitivity of 92% and a specificity of 89%, compared to the Hamilton Depression Scale. In addition, it has construct validity and concurrent predictive validity with the The International Classification of Diseases, 10th Revision (CIE-10) criteria for depression. The interpretation is made by adding the total of the first nine questions: 0-4 points, without depression; 5-9, mild depression; 10-14, moderate depression; 15-19, moderately severe depression; 20-27, severe depression.
Generalized Anxiety Disorder (GAD-7) | through study completion, an average of 2 year
  GAD-7 was originally designed primarily as a screening and severity measure for generalized anxiety disorder, this instrument also has good performance characteristics for other common anxiety disorders: panic disorder, social anxiety disorder, and post-traumatic stress disorder. This consists of 7 questions. The score is calculated by assigning scores from 0 to 3 to response categories from "Never" to "Almost Every Day." It has been validated in Spanish, where a cut-off score of 10 showed adequate values of sensitivity (86.8%) and specificity (93.4%). The scale was significantly correlated with Hamilton Anxiety scale (HAM-A) (0.852, p < 0.001), and the Hospital Anxiety and Depression Scale (HADS ) (anxiety domain, 0.903, p < 0.001). The GAD-7 total score for the seven items ranges from 0 to 21
Columbia-Suicide Severity Rating Scale (C-SSRS) | through study completion, an average of 2 year
  The first 5 items explore the presence of suicidal ideation, intention, and planning and are assessed over the past month. The sixth item explores suicidal behavior either as preparation, initiation of a suicide attempt, or a suicide attempt itself in the last three months. Each item is answered Yes or No. It has been validated in an English-speaking population (range of internal reliability goes from α=0.73 to α=0.93) and a Spanish-speaking population (α=0.53). The total score range is from 0 to 6 points. According to the answers provided To the different items, the categories of severity of suicidal ideation are established: If the answer is "Yes" to item 1 and/or item 2 and "No" to all the other items, a slight risk is indicated. If the answer is "Yes" to item 2 and answer "Yes" only to item 3, it suggests that the risk is moderate. If the answer si "Yes" to item 2 and the answer is "Yes" to any of items 4, 5, and 6, it indicates that the risk is severe.
Short Form-36 Health Survey (SF-36 v.2) | through study completion, an average of 2 year
  Instrument that assesses quality of life and general health status. It was developed by the Medical Outcome Study (MOS) and contains 36 items grouped into 8 health domains (Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health). The results of each dimension are coded and transformed into a scale ranging from 0 (the worst health status) to 100 (the best health status). Although the questionnaire is not designed to provide a global index, it allows for the calculation of two summary scores: Physical and Mental. This instrument has been validated in Chile.
Five Facet Mindfulness Questionnaire (FFMQ) | through study completion, an average of 2 year
  The original English questionnaire is a self-report of 39 items that measures Mindfulness through five facets called Observing, Describing, Acting with Awareness, Non-Judging, and Non-Reactivity. Participants must respond to each item on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true); the minimum score of the Questionnaire is 39 points and the maximum is 195 points. The instrument has adequate to good levels of reliability (Cronbach's alpha ranging from .75 to .92).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de los Andes, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Data about primary and secondary outcomes without identifiable variables such as name, date of birth, or others.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the end of the study and until five years after the end of the study.
Access Criteria: Any researchers who ask the principal investigator fot secondary analysis, data anonymized.
URL: https://www.ismeuandes.cl/

REFERENCES:
- [Background] Sheldon E, Simmonds-Buckley M, Bone C, Mascarenhas T, Chan N, Wincott M, Gleeson H, Sow K, Hind D, Barkham M. Prevalence and risk factors for mental health problems in university undergraduate students: A systematic review with meta-analysis. J Affect Disord. 2021 May 15;287:282-292. doi: 10.1016/j.jad.2021.03.054. Epub 2021 Mar 26. PMID 33812241
- [Background] Auerbach RP, Mortier P, Bruffaerts R, Alonso J, Benjet C, Cuijpers P, Demyttenaere K, Ebert DD, Green JG, Hasking P, Murray E, Nock MK, Pinder-Amaker S, Sampson NA, Stein DJ, Vilagut G, Zaslavsky AM, Kessler RC; WHO WMH-ICS Collaborators. WHO World Mental Health Surveys International College Student Project: Prevalence and distribution of mental disorders. J Abnorm Psychol. 2018 Oct;127(7):623-638. doi: 10.1037/abn0000362. Epub 2018 Sep 13. PMID 30211576
- [Background] Baader T, Rojas C, Molina JL, Gotelli M, Alamo C, Fierro C, et al. Diagnóstico de la prevalencia de trastornos de la salud mental en estudiantes universitarios y lo s factores de riesgo emocionales asociados. Revista chilena de neuro-psiquiatría. 2014;52(3):167-76.
- [Background] Barrera-Herrera A, Neira-Cofré M, Raipán-Gómez P, Riquelme-Lobos P, Escobar B. Apoyo social percibido y factores sociodemográficos en relación con los síntomas de ansiedad, depresión y estrés en universitarios chilenos. Revista de Psicopatología y Psicología Clínica. 2019;24(2).
- [Background] Hofmann SG, Gomez AF. Mindfulness-Based Interventions for Anxiety and Depression. Psychiatr Clin North Am. 2017 Dec;40(4):739-749. doi: 10.1016/j.psc.2017.08.008. Epub 2017 Sep 18. PMID 29080597
- [Background] Parcover J, Coiro MJ, Finglass E, Barr E. Effects of a brief mindfulness based group intervention on college students. Journal of college student psychotherapy. 2018;32(4):312-29.
- [Background] Demarzo M, Montero-Marin J, Puebla-Guedea M, Navarro-Gil M, Herrera-Mercadal P, Moreno-Gonzalez S, Calvo-Carrion S, Bafaluy-Franch L, Garcia-Campayo J. Efficacy of 8- and 4-Session Mindfulness-Based Interventions in a Non-clinical Population: A Controlled Study. Front Psychol. 2017 Aug 8;8:1343. doi: 10.3389/fpsyg.2017.01343. eCollection 2017. PMID 28848465
- [Background] Dimidjian S, Segal ZV. Prospects for a clinical science of mindfulness-based intervention. Am Psychol. 2015 Oct;70(7):593-620. doi: 10.1037/a0039589. PMID 26436311
- [Background] Ma L, Zhang Y, Cui Z. Mindfulness-based interventions for prevention of depressive symptoms in university students: a meta-analytic review. Mindfulness. 2019;10(11):2209-24.
- [Background] Daya Z, Hearn JH. Mindfulness interventions in medical education: A systematic review of their impact on medical student stress, depression, fatigue and burnout. Med Teach. 2018 Feb;40(2):146-153. doi: 10.1080/0142159X.2017.1394999. Epub 2017 Nov 7. PMID 29113526
- [Background] Gu J, Strauss C, Bond R, Cavanagh K. How do mindfulness-based cognitive therapy and mindfulness-based stress reduction improve mental health and wellbeing? A systematic review and meta-analysis of mediation studies. Clin Psychol Rev. 2015 Apr;37:1-12. doi: 10.1016/j.cpr.2015.01.006. Epub 2015 Jan 31. PMID 25689576
- [Background] Kabat-Zinn J. Using the wisdom of your body and mind to face stress, pain, and illness. New York, NY: Bantam Doubleday Dell. 1990;2383411.
- [Background] Williams M, Penman D. Mindfulness: a practical guide to finding peace in a frantic world: Hachette UK; 2011.
- [Background] Khoury B, Sharma M, Rush SE, Fournier C. Mindfulness-based stress reduction for healthy individuals: A meta-analysis. J Psychosom Res. 2015 Jun;78(6):519-28. doi: 10.1016/j.jpsychores.2015.03.009. Epub 2015 Mar 20. PMID 25818837
- [Background] Blanck P, Perleth S, Heidenreich T, Kroger P, Ditzen B, Bents H, Mander J. Effects of mindfulness exercises as stand-alone intervention on symptoms of anxiety and depression: Systematic review and meta-analysis. Behav Res Ther. 2018 Mar;102:25-35. doi: 10.1016/j.brat.2017.12.002. Epub 2017 Dec 20. PMID 29291584
- [Background] Godfrin KA, van Heeringen C. The effects of mindfulness-based cognitive therapy on recurrence of depressive episodes, mental health and quality of life: A randomized controlled study. Behav Res Ther. 2010 Aug;48(8):738-46. doi: 10.1016/j.brat.2010.04.006. Epub 2010 Apr 18. PMID 20462570
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Galante J, Dufour G, Vainre M, Wagner AP, Stochl J, Benton A, Lathia N, Howarth E, Jones PB. A mindfulness-based intervention to increase resilience to stress in university students (the Mindful Student Study): a pragmatic randomised controlled trial. Lancet Public Health. 2018 Feb;3(2):e72-e81. doi: 10.1016/S2468-2667(17)30231-1. Epub 2017 Dec 19. PMID 29422189
- [Background] Canby NK, Cameron IM, Calhoun AT, Buchanan GM. A brief mindfulness intervention for healthy college students and its effects on psychological distress, self-control, meta-mood, and subjective vitality. Mindfulness. 2015;6(5):1071-81.
- [Background] Cebolla A, Demarzo M, Martins P, Soler J, Garcia-Campayo J. Unwanted effects: Is there a negative side of meditation? A multicentre survey. PLoS One. 2017 Sep 5;12(9):e0183137. doi: 10.1371/journal.pone.0183137. eCollection 2017. PMID 28873417
- [Background] Segal ZV, Teasdale JD, Williams JMG. Mindfulness-Based Cognitive Therapy: Theoretical Rationale and Empirical Status. 2004.
- [Background] Segal ZV, Dimidjian S, Beck A, Boggs JM, Vanderkruik R, Metcalf CA, Gallop R, Felder JN, Levy J. Outcomes of Online Mindfulness-Based Cognitive Therapy for Patients With Residual Depressive Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Jun 1;77(6):563-573. doi: 10.1001/jamapsychiatry.2019.4693. PMID 31995132
- [Background] Querstret D, Cropley M, Fife-Schaw C. The Effects of an Online Mindfulness Intervention on Perceived Stress, Depression and Anxiety in a Non-clinical Sample: A Randomised Waitlist Control Trial. Mindfulness (N Y). 2018;9(6):1825-1836. doi: 10.1007/s12671-018-0925-0. Epub 2018 May 2. PMID 30524514
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Roberts RE, Attkisson CC, Stegner BL. A client satisfaction scale suitable for use with Hispanics? Hispanic Journal of Behavioral Sciences. 1983;5(4):461-75.
- [Background] Roberts RE, Atrkisson CC, Mendias RM. Assessing the client satisfaction questionnaire in English and Spanish. Hispanic Journal of Behavioral Sciences. 1984;6(4):385-96.
- [Background] Baader T, Molina JL, Venezian S, Rojas C, Farías R, Fierro-Freixenet C, et al. Validación y utilidad de la encuesta PHQ-9 (Patient Health Questionnaire) en el diagnóstico de depresión en pacientes usuarios de atención primaria en Chile. Revista chilena de neuro-psiquiatría. 2012;50(1):10-22.
- [Background] Garcia-Campayo J, Zamorano E, Ruiz MA, Pardo A, Perez-Paramo M, Lopez-Gomez V, Freire O, Rejas J. Cultural adaptation into Spanish of the generalized anxiety disorder-7 (GAD-7) scale as a screening tool. Health Qual Life Outcomes. 2010 Jan 20;8:8. doi: 10.1186/1477-7525-8-8. PMID 20089179
- [Background] Crockett MA, Martinez V, Ordonez-Carrasco JL. [Psychometric properties of the Generalized Anxiety Disorder 7-item (GAD-7) scale in Chilean adolescents]. Rev Med Chil. 2022 Apr;150(4):458-464. doi: 10.4067/S0034-98872022000400458. Spanish. PMID 36155755
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Schmidt C, Vinet EV. Atención plena: validación del five facet mindfulness questionnaire (FFMQ) en estudiantes universitarios chilenos. Terapia psicológica. 2015;33(2):93-102.
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Valdes JM, Diaz FJ, Christiansen PM, Lorca GA, Solorza FJ, Alvear M, Ramirez S, Nunez D, Araya R, Gaete J. Mental Health and Related Factors Among Undergraduate Students During SARS-CoV-2 Pandemic: A Cross-Sectional Study. Front Psychiatry. 2022 May 31;13:833263. doi: 10.3389/fpsyt.2022.833263. eCollection 2022. PMID 35711588
- [Background] Olivares P. Estado de Salud de Beneficiarios del Sistema de Salud de Chile, 2004-2005. Superintendencia de Isapres, Departamento de Estudios y Desarrollo; 2006.
- [Background] Breedvelt JJF, Amanvermez Y, Harrer M, Karyotaki E, Gilbody S, Bockting CLH, Cuijpers P, Ebert DD. The Effects of Meditation, Yoga, and Mindfulness on Depression, Anxiety, and Stress in Tertiary Education Students: A Meta-Analysis. Front Psychiatry. 2019 Apr 24;10:193. doi: 10.3389/fpsyt.2019.00193. eCollection 2019. PMID 31068842
- [Background] Dawson AF, Brown WW, Anderson J, Datta B, Donald JN, Hong K, Allan S, Mole TB, Jones PB, Galante J. Mindfulness-Based Interventions for University Students: A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Appl Psychol Health Well Being. 2020 Jul;12(2):384-410. doi: 10.1111/aphw.12188. Epub 2019 Nov 19. PMID 31743957
- [Background] Santorelli SF, Kabat-Zinn J, Blacker M, Meleo-Meyer F, Koerbel L. Mindfulness-based stress reduction (MBSR) authorized curriculum guide. Center for Mindfulness in Medicine, Health Care, and Society (CFM) University of Massachusetts Medical School. 2017.